CLINICAL TRIAL: NCT04484961
Title: Effects of Blood Flow Restriction Rehabilitation After Bone Patellar Tendon Bone Anterior Cruciate Ligament Reconstruction
Brief Title: Effects of Blood Flow Restriction Rehabilitation After Anterior Cruciate Ligament Reconstruction
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The Methodist Hospital Research Institute (Other)
Responsible Party: Principal Investigator, Patrick McCulloch,MD, Principal investigator, The Methodist Hospital Research Institute
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Pro000138201
Record Dates: First submitted 2020-07-13; First posted 2020-07-24 (Actual); Results first posted 2024-11-25 (Actual); Last update posted 2024-11-25 (Actual); Status verified 2024-10

CONDITIONS: ACL Tear
MeSH Terms: conditions — Anterior Cruciate Ligament Injuries | interventions — Blood Flow Restriction Therapy

STUDY DESIGN:
Intervention Model Description: Participants were randomized to either receive standard physical therapy or standard physical therapy with blood flow restriction therapy.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Control - Routine Rehab (No Intervention): Participants in this group received standard ACL rehab with no blood flow restriction therapy.
- Experimental - BFR (Experimental): Participants in this group received standard ACL rehab with the addition of blood flow restriction therapy.
  Interventions: Device: Blood flow restriction (BFR)

INTERVENTIONS:
Device: Blood flow restriction (BFR) — The study group underwent normal ACL rehab modified by use of a tourniquet for blood flow restriction during selected exercises.
  Arms: Experimental - BFR

SUMMARY:
The study is a prospective randomized control trial consisting of subjects requiring ACL reconstruction with BTB autograft. Subjects were randomly divided into two groups following their inclusion in the study. One group underwent the normal ACL rehab protocol as determined by the participating surgeons. The study group underwent normal ACL rehab modified by use of a tourniquet for blood flow restriction during selected exercises.

DETAILED DESCRIPTION:
On the day of the procedure, the surgeon will measure the subject's thigh circumference 1/3 distance from the superior pole of the patella to the inguinal crease. The subject will then undergo the normal BTB autograft ACL reconstruction procedure. A subject will be excluded from the study if a meniscal repair is performed. At the subject's two week post-operative clinic visit, the physician will measure thigh circumference at 1/3 distance from the superior pole of the patella to the inguinal crease. Study group subjects will begin physical therapy instructed BFR exercises at two weeks post operatively. Study group subjects will be taken through normal ACL rehab protocol as well as BFR exercises. Control group subjects will do the same exercises and formal physical therapy rehab protocol as the study group without BFR.

The BFR exercises will consist of: bilateral leg press week 3-10, eccentric leg press weeks 4-10, hamstring curl week 4-6, eccentric hamstring curl weeks 7-10, straight leg press weeks 6-10. The pressure used will be elevated to occluded blood flow by 80% (80% occlusion pressure) which will be determined for each individual subject. Subjects will do exercises at 20% of 1RM in 4 sets of 30-15-15-15 repetitions separated by 30 seconds of rest. Repetition maximum (1RM) will be determined by the contralateral leg, using the greatest amount of weight with full range of motion and proper form. This will be done over three separate tries, separated by one minute breaks. Resistance loads will be adjusted every 2 weeks as strength improves. During the exercise protocol, if patients are unable to complete the prescribed amount of repetitions, rest periods between sets will be increased as needed. The control group will do these exercises without BFR. Both study and control groups will also do the surgeons' standard post-ACL reconstruction physical therapy protocol.

Cuff pressures will be determined using the Loenneke et al outline, based off of thigh circumference and estimated cuff pressure for 50% artery occlusion [19].

Body composition (DEXA), bone density (DEXA), IKDC and Tegner Lysholm scores will be recorded at first rehabilitation visit, two weeks, eight weeks and 12 weeks following the initiation of rehab (1 wk following surgery). Y- balance, single leg squat distance, and single leg step down will be measured at 8 weeks and 12 weeks of rehab. Return to play will be recorded as the number of months after the day of operation until subject returns to sport.

ELIGIBILITY:
Inclusion Criteria:

* Ages 18-35
* Received ACL surgery with a patellar tendon autograft

Exclusion Criteria:

* Concomitant meniscal tear or additional ligamentous injury to the knee
* Obesity (BMI>30)
* Diabetes
* Cardiovascular, renal, liver or pulmonary disease
* Active infections
* Cancer (current or treated within the past 2 years) or coagulation disorder
* Rapid weight change within the past year
* Physically unable to participate in the intervention
* Are not currently taking, or recently (w/in 1month of participation) taken prescribed or over the counter ergogenic aids or compounds known to be banned by the NCAA. The NCAA banned substances list can be viewed from: http://www.ncaa.org/health-and-safety/policy/2014-15-ncaa-banned-drugs
* Unable to complete a minimum of 85% of the assigned rehabilitation sessions.

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 50 (Actual)
Dates: Start 2016-03-18 (Actual); Primary Completion 2020-07-10 (Actual); Study Completion 2020-07-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Patrick McCulloch, MD, Principal Investigator — The Methodist Hospital Research Institute

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Abe T, Kearns CF, Sato Y. Muscle size and strength are increased following walk training with restricted venous blood flow from the leg muscle, Kaatsu-walk training. J Appl Physiol (1985). 2006 May;100(5):1460-6. doi: 10.1152/japplphysiol.01267.2005. Epub 2005 Dec 8. PMID 16339340
- [Background] Abe T, Sakamaki M, Fujita S, Ozaki H, Sugaya M, Sato Y, Nakajima T. Effects of low-intensity walk training with restricted leg blood flow on muscle strength and aerobic capacity in older adults. J Geriatr Phys Ther. 2010 Jan-Mar;33(1):34-40. PMID 20503732
- [Background] Abe T, Yasuda T, Midorikawa T, et al. Skeletal muscle size and circulating IGF-1 are increased after two weeks of twice daily "KAATSU" resistance training. Int J KAATSU Train Res. 2005;1(1):6-12
- [Background] Anderson AW, Smith JJ. Proximal tibial fracture after patellar tendon autograft for ipsilateral ACL reconstruction. J Knee Surg. 2009 Apr;22(2):142-4. doi: 10.1055/s-0030-1247739. PMID 19476179
- [Background] Anderson MJ, Diko S, Baehr LM, Baar K, Bodine SC, Christiansen BA. Contribution of mechanical unloading to trabecular bone loss following non-invasive knee injury in mice. J Orthop Res. 2016 Oct;34(10):1680-1687. doi: 10.1002/jor.23178. Epub 2016 Feb 10. PMID 26826014
- [Background] Ardern CL, Webster KE, Taylor NF, Feller JA. Return to the preinjury level of competitive sport after anterior cruciate ligament reconstruction surgery: two-thirds of patients have not returned by 12 months after surgery. Am J Sports Med. 2011 Mar;39(3):538-43. doi: 10.1177/0363546510384798. Epub 2010 Nov 23. PMID 21098818
- [Background] Beaudart C, Dawson A, Shaw SC, Harvey NC, Kanis JA, Binkley N, Reginster JY, Chapurlat R, Chan DC, Bruyere O, Rizzoli R, Cooper C, Dennison EM; IOF-ESCEO Sarcopenia Working Group. Nutrition and physical activity in the prevention and treatment of sarcopenia: systematic review. Osteoporos Int. 2017 Jun;28(6):1817-1833. doi: 10.1007/s00198-017-3980-9. Epub 2017 Mar 1. PMID 28251287
- [Background] Bowman EN, El-shaar R, Milligan H, et al. The Proximal and Distal Effects of Blood Flow Restriction Therapy on Upper and Lower Extremity Strengthening: A Randomized Controlled Trial. Orthop J Sports Med. 2019;7(7_suppl5):2325967119S2325900337.
- [Background] Cook SB, Clark BC, Ploutz-Snyder LL. Effects of exercise load and blood-flow restriction on skeletal muscle function. Med Sci Sports Exerc. 2007 Oct;39(10):1708-13. doi: 10.1249/mss.0b013e31812383d6. PMID 17909396
- [Background] Dankel SJ, Jessee MB, Abe T, Loenneke JP. The Effects of Blood Flow Restriction on Upper-Body Musculature Located Distal and Proximal to Applied Pressure. Sports Med. 2016 Jan;46(1):23-33. doi: 10.1007/s40279-015-0407-7. PMID 26446893
- [Background] Elkasrawy M, Immel D, Wen X, Liu X, Liang LF, Hamrick MW. Immunolocalization of myostatin (GDF-8) following musculoskeletal injury and the effects of exogenous myostatin on muscle and bone healing. J Histochem Cytochem. 2012 Jan;60(1):22-30. doi: 10.1369/0022155411425389. PMID 22205678
- [Background] Fry CS, Glynn EL, Drummond MJ, Timmerman KL, Fujita S, Abe T, Dhanani S, Volpi E, Rasmussen BB. Blood flow restriction exercise stimulates mTORC1 signaling and muscle protein synthesis in older men. J Appl Physiol (1985). 2010 May;108(5):1199-209. doi: 10.1152/japplphysiol.01266.2009. Epub 2010 Feb 11. PMID 20150565
- [Background] Giles L, Webster KE, McClelland J, Cook JL. Quadriceps strengthening with and without blood flow restriction in the treatment of patellofemoral pain: a double-blind randomised trial. Br J Sports Med. 2017 Dec;51(23):1688-1694. doi: 10.1136/bjsports-2016-096329. Epub 2017 May 12. PMID 28500081
- [Background] Hamrick MW. A role for myokines in muscle-bone interactions. Exerc Sport Sci Rev. 2011 Jan;39(1):43-7. doi: 10.1097/JES.0b013e318201f601. PMID 21088601
- [Background] Korakakis V, Whiteley R, Epameinontidis K. Blood Flow Restriction induces hypoalgesia in recreationally active adult male anterior knee pain patients allowing therapeutic exercise loading. Phys Ther Sport. 2018 Jul;32:235-243. doi: 10.1016/j.ptsp.2018.05.021. Epub 2018 May 31. PMID 29879638
- [Background] Lambert B, Hedt C, Epner E, et al. BFR For Proximal Benefit: Blood Flow Restriction Therapy For The Shoulder? Med Sci Sports Exerc. 2019;51(6):972-973.
- [Background] Lambert B, Hedt CA, Jack RA, et al. Blood flow restriction therapy preserves whole limb bone and muscle following ACL reconstruction. Orthop J Sports Med. 2019;7(3_suppl2):2325967119S2325900196.
- [Background] Lambert BS, Hedt C, Moreno M, Harris JD, McCulloch P. Blood Flow Restriction Therapy for Stimulating Skeletal Muscle Growth: Practical Considerations for Maximizing Recovery in Clinical Rehabilitation Settings. Tech Orthop. 2018;33(2):89-97.
- [Background] Lambert BS, Shimkus KL, Fluckey JD, Riechman SE, Greene NP, Cardin JM, Crouse SF. Anabolic responses to acute and chronic resistance exercise are enhanced when combined with aquatic treadmill exercise. Am J Physiol Endocrinol Metab. 2015 Feb 1;308(3):E192-200. doi: 10.1152/ajpendo.00689.2013. Epub 2014 Nov 25. PMID 25425002
- [Background] Loenneke JP, Kim D, Fahs CA, Thiebaud RS, Abe T, Larson RD, Bemben DA, Bemben MG. Effects of exercise with and without different degrees of blood flow restriction on torque and muscle activation. Muscle Nerve. 2015 May;51(5):713-21. doi: 10.1002/mus.24448. PMID 25187395
- [Background] Mundermann A, Payer N, Felmet G, Riehle H. Comparison of volumetric bone mineral density in the operated and contralateral knee after anterior cruciate ligament and reconstruction: A 1-year follow-up study using peripheral quantitative computed tomography. J Orthop Res. 2015 Dec;33(12):1804-10. doi: 10.1002/jor.22962. Epub 2015 Jul 14. PMID 26123943
- [Background] Patterson SD, Brandner CR. The role of blood flow restriction training for applied practitioners: A questionnaire-based survey. J Sports Sci. 2018 Jan;36(2):123-130. doi: 10.1080/02640414.2017.1284341. Epub 2017 Feb 1. PMID 28143359
- [Background] Rosenthal R. Parametric measures of effect size. The handbook of research synthesis. 1994;621:231-244.
- [Background] Scott BR, Loenneke JP, Slattery KM, Dascombe BJ. Exercise with blood flow restriction: an updated evidence-based approach for enhanced muscular development. Sports Med. 2015 Mar;45(3):313-25. doi: 10.1007/s40279-014-0288-1. PMID 25430600
- [Background] Swift JM, Nilsson MI, Hogan HA, Sumner LR, Bloomfield SA. Simulated resistance training during hindlimb unloading abolishes disuse bone loss and maintains muscle strength. J Bone Miner Res. 2010 Mar;25(3):564-74. doi: 10.1359/jbmr.090811. PMID 19653816
- [Background] Thangamani VB, Flanigan DC, Merk BR. Intra-articular distal femur fracture extending from an expanded femoral tunnel in an anterior cruciate ligament (ACL) reconstructed knee: a case report. J Trauma. 2009 Dec;67(6):E209-12. doi: 10.1097/TA.0b013e3181469f42. PMID 19065114
- [Background] Vechin FC, Libardi CA, Conceicao MS, Damas FR, Lixandrao ME, Berton RP, Tricoli VA, Roschel HA, Cavaglieri CR, Chacon-Mikahil MP, Ugrinowitsch C. Comparisons between low-intensity resistance training with blood flow restriction and high-intensity resistance training on quadriceps muscle mass and strength in elderly. J Strength Cond Res. 2015 Apr;29(4):1071-6. doi: 10.1519/JSC.0000000000000703. PMID 25264670
- [Background] Wright R, Spindler K, Huston L, Amendola A, Andrish J, Brophy R, Carey J, Cox C, Flanigan D, Jones M, Kaeding C, Marx R, Matava M, McCarty E, Parker R, Vidal A, Wolcott M, Wolf B, Dunn W. Revision ACL reconstruction outcomes: MOON cohort. J Knee Surg. 2011 Dec;24(4):289-94. doi: 10.1055/s-0031-1292650. PMID 22303759
- [Background] Yamanaka T, Farley RS, Caputo JL. Occlusion training increases muscular strength in division IA football players. J Strength Cond Res. 2012 Sep;26(9):2523-9. doi: 10.1519/JSC.0b013e31823f2b0e. PMID 22105051
- [Background] Zargi T, Drobnic M, Strazar K, Kacin A. Short-Term Preconditioning With Blood Flow Restricted Exercise Preserves Quadriceps Muscle Endurance in Patients After Anterior Cruciate Ligament Reconstruction. Front Physiol. 2018 Aug 24;9:1150. doi: 10.3389/fphys.2018.01150. eCollection 2018. PMID 30197599

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Houston hospital and clinic locations
Pre-assignment Details: Examples of why a patient might be enrolled and then not assigned to a study arm would be:
  * new injury
  * deciding on a different PT location
  * time constraints
Period: Overall Study
Arm/Group | Control - Routine Rehab | Experimental - BFR
Started | 24 | 26
Completed | 15 | 17
Not Completed | 9 | 9
Not completed — Lost to Follow-up | 9 | 9

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Control - Routine Rehab | Experimental - BFR | Total
Number analyzed (Participants) | 24 | 26 | 50
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 24 | 26 | 50
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11 | 8 | 19
  Male | 13 | 18 | 31
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.

OUTCOME MEASURES:

1. Primary Outcome: Determine if BFR Changes Loss of LE Lean Muscle Mass
Description: LE lean muscle mass was measured in kilograms using DEXA (iDXA, GE®)
Time Frame: Pre-surgery, 6 weeks post-surgery and 12 weeks post-surgery
Measure: Mean (Standard Deviation); unit: kg
Groups:
- Control: Standard PT, No BFR Injured Limb
- Experimental - BFR: Standard PT, BFR Injured Limb
Arm/Group | Control | Experimental - BFR
Number analyzed (Participants) | 15 | 17
kg
  Pre-Surgery Whole Limb Lean Mass | 8.97 (0.21) | 8.97 (0.20)
  6 week post surgery Whole Limb Lean Mass | 8.37 (0.21) | 8.93 (0.20)
  12 Week Post Surgery Whole Limb Lean Mass | 8.58 (0.21) | 9.04 (0.20)
  Pre-Surgery Thigh Lean Mass | 3.18 (0.07) | 3.18 (0.06)
  6 week post surgery Thigh Lean Mass | 2.91 (0.07) | 3.10 (0.06)
  12 week post surgery Thigh Lean Mass | 3.04 (0.07) | 3.18 (0.06)

2. Primary Outcome: Determine if BFR Changes Loss of Bone Mass
Description: Bone mass was measured in grams using DEXA (iDXA, GE®)
Time Frame: Pre-surgery, 6 weeks post-surgery and 12 weeks post-surgery
Measure: Mean (Standard Deviation); unit: g
Arm/Group | Control | Experimental - BFR
Number analyzed (Participants) | 15 | 17
g
  Whole Limb Bone Mass at Pre-surgery | 567.9 (6.4) | 568.2 (6.1)
  Whole Limb Bone Mass at 6 weeks post-operation | 555 (6.4) | 567.2 (6.1)
  Whole Limb Bone Mass at 12 weeks post-operation | 550.9 (6.4) | 565.4 (6.1)
  Femur Bone Mass at Pre-surgery | 156.2 (2.5) | 156.4 (2.3)
  Femur Bone Mass at 6 weeks post surgery | 151.2 (2.5) | 154.3 (2.3)
  Femur Bone Mass at 12 weeks post surgery | 148.9 (1.8) | 153 (1.7)

3. Primary Outcome: Determine if BFR Changes Loss of Bone Mineral Density
Description: Bone mineral density was measured in grams/cm2 using DEXA (iDXA, GE®)
Time Frame: Pre-surgery, 6 weeks post-surgery and 12 weeks post-surgery
Measure: Mean (Standard Deviation); unit: g/cm^2
Arm/Group | Control | Experimental - BFR
Number analyzed (Participants) | 15 | 17
g/cm^2
  Distal Femur Bone Mineral density at pre-surgery | 1.2 (0.02) | 1.2 (0.02)
  Distal Femur Bone Mineral density at 6 weeks post-operation | 1.1 (0.02) | 1.2 (0.02)
  Distal Femur Bone Mineral density at 12 weeks post-operation | 1.1 (0.02) | 1.1 (0.02)
  Proximal Tibia Bone Mineral density at pre-surgery | 1.47 (0.02) | 1.47 (0.04)
  Proximal Tibia Bone Mineral density at 6 weeks post surgery | 1.40 (0.02) | 1.44 (0.04)
  Proximal Tibia Bone Mineral density at 12 weeks post surgery | 1.35 (0.03) | 1.44 (0.03)
  Proximal Fibia Bone Mineral Density at pre-surgery | 0.46 (0.02) | 0.46 (0.02)
  Proximal Fibia Bone Mineral Density at 6 weeks post-surgery | 0.40 (0.02) | 0.42 (0.02)
  Proximal Fibia Bone Mineral Density at 12 weeks post surgery | 0.38 (0.02) | 0.43 (0.02)

4. Secondary Outcome: Does BFR Change the Number of Exercise Repetitions in Functional Physical Therapy Testing
Description: Single leg (SL) squat (best of 3 attempts)
Time Frame: Week 8 and Week 12 post-surgery
Measure: Mean (Standard Deviation); unit: cm
Arm/Group | Control | Experimental - BFR
Number analyzed (Participants) | 15 | 17
cm
  SL Squat Week 8 | 34.3 (6.3) | 33.4 (5.1)
  SL Squat Week 12 | 40.9 (5.4) | 43.0 (5.5)

5. Secondary Outcome: Does BFR Change the Number of Exercise Repetitions in Functional Physical Therapy Testing
Description: SL eccentric step down (reps to fatigue or inadequate technique)
Time Frame: 8 weeks post surgery, 12 weeks post surgery
Measure: Mean (Standard Deviation); unit: reps
Arm/Group | Control | Experimental - BFR
Number analyzed (Participants) | 15 | 17
reps
  SL eccentric step down at 8 weeks post surgery | 44.3 (14.7) | 45.1 (13.9)
  SL eccentric step down at 12 weeks post surgery | 61.0 (18.6) | 62.7 (18.0)

6. Secondary Outcome: Does BFR Change the Number of Exercise Repetitions in Functional Physical Therapy Testing
Description: Y-balance anterior (best of 3 attempts)
Time Frame: 8 weeks post surgery, 12 weeks post surgery
Measure: Mean (Standard Deviation); unit: cm
Arm/Group | Control | Experimental - BFR
Number analyzed (Participants) | 15 | 17
cm
  Y-balance anterior (best of 3 attempts) at 8 weeks post surgery | 48.7 (14.3) | 50.0 (2.2)
  Y-balance anterior (best of 3 attempts) at 12 weeks post surgery | 55.9 (18.6) | 62.7 (18.0)

7. Secondary Outcome: Does BFR Change the Number of Exercise Repetitions in Functional Physical Therapy Testing
Description: Y-balance posteromedial (best of 3 attempts)
Time Frame: 8 weeks post surgery, 12 weeks post surgery
Measure: Mean (Standard Deviation); unit: cm
Arm/Group | Control | Experimental - BFR
Number analyzed (Participants) | 15 | 17
cm
  Y-balance posteromedial (best of 3 attempts) at 8 weeks post surgery | 93.3 (8.6) | 93.9 (7.4)
  Y-balance posteromedial (best of 3 attempts) at 12 weeks post surgery | 104.4 (9.2) | 100.0 (8.5)

8. Secondary Outcome: Does BFR Change the Number of Exercise Repetitions in Functional Physical Therapy Testing
Description: Y-balance posterolateral (best of 3 attempts)
Time Frame: 8 weeks post surgery, 12 weeks post surgery
Measure: Mean (Standard Deviation); unit: cm
Arm/Group | Control | Experimental - BFR
Number analyzed (Participants) | 15 | 17
cm
  Y-balance posterolateral (best of 3 attempts) at 8 weeks post surgery | 90.3 (10.3) | 91.9 (4.6)
  Y-balance posterolateral (best of 3 attempts) at 12 weeks post surgery | 104.5 (9.2) | 99.7 (8.5)

9. Secondary Outcome: Does BFR Change the Number of Exercise Repetitions in Functional Physical Therapy Testing
Description: SL leg press (1RM)
Time Frame: 8 weeks post surgery, 12 weeks post surgery
Measure: Mean (Standard Deviation); unit: kg
Arm/Group | Control | Experimental - BFR
Number analyzed (Participants) | 15 | 17
kg
  SL leg press (1RM) at 8 weeks post surgery | 58.6 (8.0) | 59.3 (10.0)
  SL leg press (1RM) at 12 weeks post surgery | 76.5 (9.0) | 72.7 (8.7)

10. Secondary Outcome: Does BFR Change the Number of Exercise Repetitions in Functional Physical Therapy Testing
Description: SL hamstring curl (1RM)
Time Frame: 8 weeks post surgery, 12 weeks post surgery
Measure: Mean (Standard Deviation); unit: kg
Arm/Group | Control | Experimental - BFR
Number analyzed (Participants) | 15 | 17
kg
  SL hamstring curl (1RM) at 8 weeks post surgery | 29.9 (5.1) | 28.2 (4.2)
  SL hamstring curl (1RM) at 12 weeks post surgery | 38.5 (4.5) | 37.7 (4.9)

ADVERSE EVENTS:
Time Frame: 12 weeks after surgery
Groups:
- Treatment Group: BFR: BFR Treatment Group
- Control - Routine Rehab: Control Group
Arm/Group | Treatment Group: BFR | Control - Routine Rehab
All-Cause Mortality (participants affected / at risk) | 0/26 | 0/24
Serious Adverse Events (participants affected / at risk) | 0/26 | 0/24
Other Adverse Events (participants affected / at risk) | 1/26 | 0/24
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment Group: BFR (N=26) | Control - Routine Rehab (N=24)
Mild Muscle Strain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) — The subject had a mild muscle strain at the 12 week mark. This was a single episode treated with ibuprofen per the PI.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol (2015-12-28): https://cdn.clinicaltrials.gov/large-docs/61/NCT04484961/Prot_000.pdf